CLINICAL TRIAL: NCT06061939
Title: Effects of a Resistance Training Program Based on Blood Flow Restriction Training for People Over 45 Years of Age With Multiple Sclerosis on Muscle Strength and Functionality.
Brief Title: Effects of Blood Flow Restriction Training on Middle-aged People With Multiple Sclerosis.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Jaén (Other)
Responsible Party: Principal Investigator, Agustín Aibar Almazán, Principal investigator, University of Jaén
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: University of Jaén*
Record Dates: First submitted 2023-09-25; First posted 2023-09-29 (Actual); Last update posted 2025-05-30 (Actual); Status verified 2025-05

CONDITIONS: Sclerosis, Multiple
MeSH Terms: conditions — Multiple Sclerosis | interventions — Blood Flow Restriction Therapy

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (No Intervention): A control group (CG) that will not undergo treatment, which will be evaluated in the pre and post phase of the study. Participants assigned to this group will receive general advice on the positive effects of regular physical activity, and they will be given the guide of recommendations for the promotion of physical activity.
- Intervention Group (Experimental): An experimental group (EG) that after an initial evaluation and with their consent, will be subjected to a directed physical training program, based on strength training with blood flow restriction, applied for 12 weeks with 3 weekly sessions (Monday, Wednesday and Friday), with a duration of 30-45 minutes per session. The exercises to be performed will be divided into three different phases: warm-up during the first 10 minutes; the main part with a duration of 15 minutes (where each exercise must be performed doing 4 series with a pattern of 30-15-15-15 repetitions, resting 30-45 seconds between series and 1-2 minutes between exercises); and the return to calm, based above all on stretching exercises with a total duration of 10 minutes.
  Interventions: Other: Blood Flow Restriction training with Oclussion Cuff.

INTERVENTIONS:
Other: Blood Flow Restriction training with Oclussion Cuff. — A strength training program with blood flow restriction will be performed for 12 weeks, with 30-45 minute sessions on Mondays, Wednesdays and Fridays. Each session includes a warm-up, the main part with specific exercises and a cool-down with stretching.
  Arms: Intervention Group

SUMMARY:
To analyze the effects of a resistance training program based on the blood flow restriction modality on muscle strengthening and functionality in people over 45 years of age with multiple sclerosis (MS).

DETAILED DESCRIPTION:
This research corresponds to an experimental study, a double-blind randomized controlled clinical trial, where a total of blood flow (n = X) 12 weeks; and the control group (n= X) that will only receive general recommendations about the benefits of physical exercise. The variables will be measured for both groups with the same validated tools and the same researcher to avoid information bias and differential misclassification. The evaluations will be carried out at the beginning of the intervention and immediately after the end of this period, and the results will be noted in a data record that will later be unified in an Excel database, registering a code for each participant to maintain condition. of privacy, but at the same time allow the required comparability.

For the independent variables, sociodemographic characteristics, clinical history and the socio-familial assessment scale will be addressed; For their part, the result variables are divided by areas: those focused on the health status of patients with MS will measure the level of disability through the Expanded Disability Status Scale (EDSS), the impact of MS through the Multiple Sclerosis Impact Scale 29 (MSIS-29) and health-related quality of life (HRQoL) with the Short Form-36 (SF-36). For the physical condition variables, the Maximal Voluntary Isometric Contraction (MVIC) will be used with a dynamometer to measure general muscle strength and grip strength, as well as the Sit to Stand-5 repetitions (STS-5) and the Sit to Stand-5 repetitions (STS-5). 30 seconds (STS-30) to evaluate lower limb strength. For the functional variables, the impact on walking is evaluated using the Timed 25-Foot Walking Test (T25FWT); gait speed with the 10-Meters Walk Test (10-MWT) and Timed Up and Go (TUG); while walking endurance will be measured with the 6-Minute Walk Test (6-MWT). For its part, postural stability and balance from the Berg Balance Scale (BBS). To evaluate the level of physical activity, Godin Leisure-Time Exercise Questionnaire scores (GLTEQ) will be used. The questionnaire to determine fatigue will be the Fatigue Severity Scale (FSS) and the one in charge of measuring cognitive function will be the Symbol Digit Modalities Test (SDMT). On the other hand, in the psychological variables, the Hospital Anxiety and Depression Scale (HADS) will be applied for anxiety and depression and the Perceived Stress Scale (PSS) for the stress level. Finally, to measure sleep quality, the Pittsburgh Sleep Quality Index (PSQI) will be used. All variables will have pre and post intervention measurements. As a result, a training program with blood flow restriction is expected to improve the health status, muscle strength, functionality and psychological domains of middle-aged patients (> 45 years) with MS, thus contributing to the comprehensive approach of this population. Once the intervention is completed, the final evaluation will be carried out and, based on the comparative process, define whether there are significant differences with respect to the results initially obtained.

ELIGIBILITY:
Inclusion Criteria:

* Male and female users over 45 years of age, who voluntarily agree to participate in the study, who are able to understand the instructions and exercise protocols of this project.

Exclusion Criteria:

* People with contraindications for performing physical tests or exercise. Users with a diagnosis of pathologies such as cancer, pulmonary hypertension and kidney failure, population with a diagnosis of heart disease or heart failure, population with a diagnosis and/or under psychiatric management, with neurological or cognitive alterations will be excluded. Population diagnosed with Human Immunodeficiency Virus infection or disease (HIV/AIDS). Population that does not agree to participate in the study or who, at the time of entering the program, have denied the endorsement of the use of their data for research in the informed consent.

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 94 (Actual)
Dates: Start 2024-03-05 (Actual); Primary Completion 2024-03-11 (Actual); Study Completion 2024-06-07 (Actual)

PRIMARY OUTCOMES:
Disability Status | Up to twelve weeks
  Expanded Disability Status Scale (EDSS). Method to quantify disability in multiple sclerosis and monitor changes in the level of disability over time. It is widely used in clinical trials and in the evaluation of people with MS. The EDSS scale ranges from 0 to 10 units with 0.5 point increments representing higher levels of disability. The first levels 1.0 to 4.5 refer to people with a high degree of ambulatory capacity and the later levels 5.0 to 9.5 refer to the loss of ambulatory capacity.
Multiple Sclerosis Impact | Up to twelve weeks
  Multiple Sclerosis Impact Scale 29 (MSIS-29). It is a 29-item, condition-specific self-report questionnaire to measure the impact of MS on people's lives. It has two subscales: a 20-item physical impact scale and a 9-item psychological impact scale. It is currently in its second version, which has four-point response categories for each item: "not at all," "a little," "moderately," and "extremely." The physical impact scale can range from 20 to 80 and the psychological impact scale from 9 to 36, with lower scores indicating little impact of MS and higher scores indicating greater impact.
Short Form-36 (SF-36). | Up to twelve weeks
  It is the most used scale for the general evaluation of health-related quality of life and consists of 36 items that are grouped into eight subscales or domains: (i) physical functioning (ten items); (ii) physical role (four items); (iii) body pain (two items); (iv) general health (five articles); (v) vitality (four items); (vi) social functioning (two items); (vii) emotional role (three items); and (viii) mental health (five items). The SF-36 also provides summary assessment for the physical and mental components (PCS and MCS, respectively). Higher scores reveal better overall HRQoL.
Muscle strength | Up to twelve weeks
  Maximal Voluntary Isometric Contraction (MVIC) with the use of a dynamometer, a standardized method to measure muscle strength in patients with neuromuscular diseases5. Sit to Stand-5 repetitions (STS-5) along with Sit to Stand-30 seconds (STS-30) for MMII strength. In these tests, the patient must get up from a chair and measure the time it takes to perform 5 repetitions or quantify the number of repetitions that the patient is able to perform in 30 seconds6,7. For STS-5 the cut-off point is set at 9.4 sec. for those under 60 years of age; 11.4 sec. between 60 to 69 years old; 12.6 sec. 70 to 79 years and 14.9 sec. between 80 to 89 years, below these values there would be muscle dysfunction8. In the STS-30, scores lower than 8 repetitions imply muscle dysfunction.
Gait impact | Up to twelve weeks
  Timed 25-Foot Walking Test (T25FWT). It consists of measuring the time required to travel a distance of 25 feet (7.5 meters). A time below 6 seconds means a functional gait, between 6 and 7.99 seconds means moderate gait dysfunction and 8 seconds or more means gait dysfunction.
Anxiety and depression | Up to twelve weeks
  Hospital Anxiety and Depression Scale (HADS). This scale consists of 14 items with 4 response alternatives ranging from 0 to 3 for a total of 0 to 21 points. It has 2 subscales and the score is obtained by adding the scores of each item that make it up, the interpretation criteria being the following: Range of normality (0-7), Possible case of anxiety or depression (8-10) and Case of anxiety or depression (11-21).
Sleep quality | Up to twelve weeks
  Pittsburgh Sleep Quality Index (PSQI). The PSQI consists of 19 self-assessment questions or items and 5 more to be completed by the person with whom the participant shares a bed or room (although the latter is only used to provide clinical information). These items generate a total score and 7 components or domains: sleep quality; sleep latency; sleep duration; sleep efficiency; sleep disorders; use of sleeping medications; daytime dysfunction. The PSQI total score ranges from 0 to 21, with a higher score indicating poorer sleep quality.
Walking speed | Up to twelve weeks
  10-Meters Walk Test (10-MWT) and Timed Up and Go (TUG). 10-MWT is used to measure walking speed and consists of measuring the time taken to travel 10 meters of distance11. The cut-off point is set by the walking speed in m/s, so there is no gait limitation if the speed is <0.40 m/s; moderate limitation if 0.40 to <0.80 m/s; and gait limitation ≥0.80 m/s12. On the other hand, the TUG consists of measuring the time it takes for the person to get up from a chair, walk 3 meters at their usual pace, turn around, return to the chair and sit down. 2 attempts are made and the best time is chosen. It is considered low risk of falling if the time is < 10 seconds, slight risk of falling if the time is between 10-20 seconds, and high risk of falling if the time is > 20 seconds.
Physical fitness | Up to twelve weeks
  Godin Leisure-Time Exercise Questionnaire (GLTEQ). This questionnaire consists of 3 items divided according to the intensity of the exercises performed. For each item, a score is added based on the participant's response. The scores of the items will be added, considering that the physical activity carried out is Intense ≥ 24 units, Moderate ≥14 and ≤23 units and Light < 14 units.
Walking endurance | Up to twelve weeks
  6-Minute Walk Test (6-MWT). Test commonly used for the objective evaluation of functional exercise capacity. The patient is asked to walk (minimum in a 30 meter hallway) for a period of 6 minutes, with the primary outcome measure being the distance walked in 6 minutes measured in meters. In general, normal ranges are between 400-700 meters, with a value below 400 meters being an indicator of low aerobic capacity and good above 700 meters.
Balance and gait | Up to twelve weeks
  Tinetti. Completion time: 8-10 minutes. While walking behind the patient, the evaluator asks them to respond to the questions from the gait subscale. To answer the balance subscale, the interviewer stands next to the patient. A higher score indicates better functioning. The maximum score for the gait subscale is 12, and for the balance subscale, it is 16. The sum of both scores is used to assess the risk of falls. A higher score indicates a lower risk. A score of less than 19 signifies a high risk of falls.
Multiple Sclerosis Quality of Life-54 | Up to twelve weeks
  There is no single overall score for the MSQOL-54. Two summary scores - physical health and mental health - can be derived from a weighted combination of scale scores. In addition, there are 12 subscales: physical function, role limitations-physical, role limitations-emotional, pain, emotional well-being, energy, health perceptions, social function, cognitive function, health distress, overall quality of life, and sexual function. There are also two single-item measures: satisfaction with sexual function and change in health.
Executive functions | Up to twelve weeks
  The Trail Making Test (TMT) will be used for the assessment of executive function and specifically measures timed visual and motor tasks. This test is divided into two parts: part A (TMT-A) is responsible for evaluating psychomotor attention and speed and consists of connecting consecutively numbered circles; and Part B (TMT-B), which is based on connecting alternating circles of letters and numbers and measures executive function. A longer time spent completing the test is interpreted as worse performance.
Fatigue | Up to twelve weeks
  Fatigue Severity Scale (FSS). One of the most widely used self-report tools to assess fatigue. It is made up of nine elements (1 to 7). The average score of the nine items is used as the total score of the FSS. A higher score indicates greater severity of fatigue. MID ranges from 0.5 to 1.2 for FSS total score.

SECONDARY OUTCOMES:
Symbol Digit Modalities Test (SDMT) | Up to twelve weeks
  This test measures processing speed. The SDMT sheet consists of a header with a key that relates the numbers 1 to 9 with different symbols. Below is a template with several symbols that must be assigned the corresponding number. The patient completes the first ten boxes to familiarize himself and then has 90 seconds to complete the greatest number of boxes. 44 is considered the cut-off point, so scores below 44 imply abnormal cognitive functioning, with 44 points onwards being normal.
Stress level | Up to twelve weeks
  Perceived Stress Scale (PSS). This scale is a self-report instrument that evaluates the level of perceived stress during the last month, it consists of 14 items with a response format of a five-point scale (0 = never, 1 = almost never, 2 = occasionally when, 3 = often, 4 = very often). The total score of the PSS is obtained by reversing the scores of items 4, 5, 6, 7, 9, 10 and 13 (in the following sense: 0=4, 1=3, 2=2, 3=1 and 4 =0) and then adding the 14 items. The direct score obtained indicates that a higher score corresponds to a higher level of perceived stress.
MoCA (Montreal Cognitive Assessment) | Up to twelve weeks
  Instrument that examines the skills of attention, concentration, executive functions, memory, language, visuoconstructive abilities, calculation and orientation and the maximum score is 30.
Mini-Mental State Examination (MMSE) | Up to twelve weeks
  The most widely used cognitive screening test to assess suspected symptoms consistent with cognitive impairment or dementia. Written test with a maximum score of 30. The cut-off point established for the MMSE defines "normal" cognitive function is generally set at 24, lower scores indicate more serious cognitive problems.
Chair sit and reach test | Up to twelve weeks
  To test low back and hamstring flexibility.
Back scratch test | Up to twelve weeks
  To measure general shoulder range of motion.
Isaacs Test. | Up to twelve weeks
  This test measures verbal fluency. The patient is asked to name as many elements as she can remember from each of the 4 categories: colors, animals, fruits and cities. One point is awarded for each correct item, with a maximum of 10 scoring items in each set. The patient has a maximum of 1 minute per category. Repetitions or names that do not belong to the requested category do not score, although it is useful to note the number of such cases. Always write down the names that the patient mentions, as this will help in evaluating the patient's progress. The score ranges between 0 and 40 points. The cut-off point for detecting dementia, in the Spanish validation, is equal to or less than 29 in adults, and equal to or less than 27 in older people. Furthermore, a cut-off point of 25 is proposed to consider probable Alzheimer's dementia, with a sensitivity of 87% and a specificity of 67%, resulting in a misclassification rate of 24%.
Stoicism | Up to twelve weeks
  Liverpool Stoicism Scale. The LSS is a self-reported questionnaire designed to measure stoicism; it consists of 20 items whose content refers to lack of emotional involvement, dislike for openly expressing emotion, and the ability to withstand emotion. Responses were recorded on a 5-point Likert scale ranging from strongly disagree to strongly agree. To prevent response bias, half of the questions were posed in such a way that agreement was synonymous with high stoicism, whereas for the other half, disagreement indicated a high level of stoicism. The answers to these questions were evaluated in reverse. Ten items (1, 2, 5, 7, 9, 12, 13, 15, 17, and 18) are reverse-scored. The minimum sum score is 20 and the maximum is 100. Higher scores indicate greater stoicism levels. The original version is reported to have acceptable internal consistency.
Hand coordination | Up to twelve weeks
  9 Hole Peg Test. The Nine Hole Peg Test is a simple and quick assessment tool that we occupational therapists use to evaluate manipulative dexterity, eye-hand coordination, and other upper limb functions in people with neurological impairments. It involves placing and removing nine pegs in the shortest possible time. The shorter the time, the better the score.

CONTACTS AND LOCATIONS:
Locations (1):
- Asociación Jiennense de Esclerosis Múltiple, Jaén, Spain

IPD SHARING:
Plan to Share IPD: No